CLINICAL TRIAL: NCT01178710
Title: The Cardiac Protective Effect of Simvastatin on Cardiac Surgery: a Double Blind, Randomised Clinical Trial
Brief Title: Effect of Simvastatin on Cardiac Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jing-song Ou, associate chief, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: statinstudy1
Record Dates: First submitted 2010-08-09; First posted 2010-08-10 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Rheumatic Heart Disease; Congenital Heart Disease; Aneurysm; Heart Valve Disease
MeSH Terms: conditions — Rheumatic Heart Disease; Heart Defects, Congenital; Aneurysm; Heart Valve Diseases | interventions — Simvastatin; Simcor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treatment (Experimental)
  Interventions: Drug: Simvastatin
- untreated (No Intervention): control

INTERVENTIONS:
Drug: Simvastatin — 20 mg per day, start at 5 days before surgery and continue for one year. For some congenital heart diseases which other drugs such as digoxin, antistone, furosemide were prescribed less than half year, simvastatin will be prescribed less than half year.
  Other Names: simcor
  Arms: treatment

SUMMARY:
It is well know that statins have been used to low cholesterol to prevent and treat coronary artery disease for many years. It was also reported that statins could protect endothelial function and cardiac function during coronary artery bypass graft. However, some results were controversial. Also, there is no clinical data available on statin cardiac protection during surgery in China where rheumatic heart disease is prevalent. Thus, the investigators are trying to see whether statins can protect heart injury during cardiac surgery in Chinese. Part of patients will receive statin treatment and part of will not before surgery in the study. Both patients' heart function will be measured and compared after surgery to determine whether statins can protect heart injury during heart surgery.

DETAILED DESCRIPTION:
Cardiac function is crucial for cardiac surgery. The mortality remains very high in patients with poor cardiac function preoperation, long surgical time, complicate or difficult surgical procedure or uncompleted corrected malformation currently. Thus, it is necessary to search other approaches to improve cardiac function for cardiac surgery patients in order to increase the success, decrease complication and mortality in cardiac surgery.

Although statin has been used to low cholesterol to prevent and treat coronary artery disease for many years, it has been reported that statin could protect endothelial function and cardiac function in coronary artery bypass graft. However, some results were controversy. Also, there is no clinical data available on statin cardiac protection during surgery in China where rheumatic heart disease is prevalence.Thus, it is necessary to perform a double blind, randomised clinical trial in China to determine whether statin can protect heart injury during heart surgery in China and what's its mechanism.

ELIGIBILITY:
Inclusion Criteria:

* cyanotic congenital heart disease
* noncyanotic congenital heart disease with pulmonary hypertension
* Heart valve disease,
* other heart and great artery diseases need heart or great artery surgery

Exclusion Criteria:

* Coronary artery disease
* under 10-year-old.
* noncyanotic congenital heart disease without pulmonary hypertension
* poor liver function such AST elevated,Hepatitis
* Gestation women and Breast-feeding women

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
plasma troponin T level | within the first 7 days after surgery
  The investigator will measure the plasma troponin T level in several time points before and after surgery in each patient.

SECONDARY OUTCOMES:
the index of B ultrasound on heart | one year after surgery
  Each patient will be followed up and checked with B ultrasound on heart in 1,3,6 and 12 months after surgery. The index of B ultrasound on heart, such as ejection fraction, the diameter of left ventricle, will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Jing-song Ou, MD,PhD, Principal Investigator — The Frist Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Result] White CW, Gobel FL, Campeau L, Knatterud GL, Forman SA, Forrester JS, Geller NL, Herd JA, Hickey A, Hoogwerf BJ, Hunninghake DB, Rosenberg Y, Terrin ML; Post Coronary Artery Bypass Graft Trial Investigators. Effect of an aggressive lipid-lowering strategy on progression of atherosclerosis in the left main coronary artery from patients in the post coronary artery bypass graft trial. Circulation. 2001 Nov 27;104(22):2660-5. doi: 10.1161/hc4701.099730. PMID 11723015
- [Result] Ali IS, Buth KJ. Preoperative statin use and outcomes following cardiac surgery. Int J Cardiol. 2005 Aug 3;103(1):12-8. doi: 10.1016/j.ijcard.2004.06.006. Epub 2004 Nov 6. PMID 16061117
- [Result] Greer JJ, Kakkar AK, Elrod JW, Watson LJ, Jones SP, Lefer DJ. Low-dose simvastatin improves survival and ventricular function via eNOS in congestive heart failure. Am J Physiol Heart Circ Physiol. 2006 Dec;291(6):H2743-51. doi: 10.1152/ajpheart.00347.2006. Epub 2006 Jul 14. PMID 16844920
- [Derived] Almansob MA, Xu B, Zhou L, Hu XX, Chen W, Chang FJ, Ci HB, Yao JP, Xu YQ, Yao FJ, Liu DH, Zhang WB, Tang BY, Wang ZP, Ou JS. Simvastatin reduces myocardial injury undergoing noncoronary artery cardiac surgery: a randomized controlled trial. Arterioscler Thromb Vasc Biol. 2012 Sep;32(9):2304-13. doi: 10.1161/ATVBAHA.112.252098. Epub 2012 Jul 12. PMID 22796581
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/